CLINICAL TRIAL: NCT05357105
Title: Rebound Pain Following Surgery With Regional Anesthesia Block: A Prospective Cohort Study
Brief Title: Rebound Pain Following Surgery With Regional Anesthesia Block
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: ReboundPain
Record Dates: First submitted 2022-01-14; First posted 2022-05-02 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Regional Anesthesia Morbidity; Pain, Postoperative
Keywords: Rebound Pain; Nerve Block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Regional Nerve Block Patients: Patients who receive regional nerve blocks as part of the anesthetic management prior to surgery.
  Interventions: Other: Numerical Pain Scales

INTERVENTIONS:
Other: Numerical Pain Scales — Patients who are about to receive regional nerve blocks will be administered a numerical pain scale (NRS) before, during and after the offset of the nerve block.

SUMMARY:
For some kinds of surgery, Anesthesiologists provide nerve blocks (regional anesthesia) to reduce pain from surgery by injecting freezing medication around deep nerves with ultrasound. Nerve blocks help with pain control following surgery and reduce the amount of strong opioids needed but relatively little research has focused on the pain that occurs once the nerve block has worn off. This is called rebound or transition pain.

This research study will prospectively collect data including pain scores before, during and after nerve blocks are given for surgery. We will look at the type of nerve blocks and other analgesia medications used with the aim of quantifying rebound pain to better understand how to limit it's impact on quality postoperative pain control.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Receiving peripheral nerve block as part for anesthesia/analgesia as part of standard perioperative care for surgery performed at University of Alberta Hospital during a 6 month period
* Elective and emergency surgery

Exclusion Criteria:

* Inability to consent to participate in the study (illiteracy, <7th grade education)
* Contraindication/history of hypersensitivity to local anesthetics

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients 18-75 years who are receiving peripheral nerve block as part for anesthesia/analgesia as part of standard perioperative care for surgery performed at University of Alberta Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Scale | 2-3 times per patient over the course of a nerve block, up to 48 hours after the stop of the block (single shot or cessation of nerve catheter)

CONTACTS AND LOCATIONS:
Overall Officials: James Green, MD, Principal Investigator — University of Alberta Department of Anesthesiology and Pain Medicine
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koepke EJ, Manning EL, Miller TE, Ganesh A, Williams DGA, Manning MW. The rising tide of opioid use and abuse: the role of the anesthesiologist. Perioper Med (Lond). 2018 Jul 3;7:16. doi: 10.1186/s13741-018-0097-4. eCollection 2018. PMID 29988696
- [Background] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Background] Sunderland S, Yarnold CH, Head SJ, Osborn JA, Purssell A, Peel JK, Schwarz SK. Regional Versus General Anesthesia and the Incidence of Unplanned Health Care Resource Utilization for Postoperative Pain After Wrist Fracture Surgery: Results From a Retrospective Quality Improvement Project. Reg Anesth Pain Med. 2016 Jan-Feb;41(1):22-7. doi: 10.1097/AAP.0000000000000325. PMID 26650425
- [Background] Lavand'homme P. Rebound pain after regional anesthesia in the ambulatory patient. Curr Opin Anaesthesiol. 2018 Dec;31(6):679-684. doi: 10.1097/ACO.0000000000000651. PMID 30124544
- [Background] Barry GS, Bailey JG, Sardinha J, Brousseau P, Uppal V. Factors associated with rebound pain after peripheral nerve block for ambulatory surgery. Br J Anaesth. 2021 Apr;126(4):862-871. doi: 10.1016/j.bja.2020.10.035. Epub 2020 Dec 31. PMID 33390261